CLINICAL TRIAL: NCT03014752
Title: Comparison of the Effectiveness of the Outpatient Classical Ketogenic Diet and Modified Atkins Diet on Seizures Frequency, Nutritional Status and Some Biochemical Factors in Children and Adolescents With Intractable Epilepsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9311468002
Record Dates: First submitted 2016-12-31; First posted 2017-01-09 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2016-12

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Classical ketogenic diet (Active Comparator): The classical ketogenic diet with 4:1 ketogenic ratio, each 4 grams of fat to each gram of carbohydrate plus protein, will be introduced.
  Interventions: Other: Classical ketogenic diet
- Modified Atkins diet (Active Comparator): The modified Atkins diet with a ratio of 1 or 2 to 1 (1:1, 2:1), each 1 or 2 grams of fat to each gram of carbohydrate plus protein, will be introduced gradually.
  Interventions: Other: Modified Atkins diet

INTERVENTIONS:
Other: Classical ketogenic diet — The classical ketogenic diet with a ratio of 4 to 1 (4:1), each 4 grams of fat to each gram of carbohydrate plus protein, will be introduced gradually.
  Arms: Classical ketogenic diet
Other: Modified Atkins diet — The modified Atkins diet with a ratio of 1 or 2 to 1 (1:1, 2:1), each 1 or 2 grams of fat to each gram of carbohydrate plus protein, will be introduced gradually.
  Other Names: MAD
  Arms: Modified Atkins diet

SUMMARY:
Epilepsy is one of a common neurological disorder. Antiepileptic drugs (AEDs) are usually the primary treatment of epilepsy. However, almost 30% of patients do not respond to AEDs and other treatments including ketogenic diet (KD) are used. The Ketogenic Diet (KD) is a low-carbohydrate, high fat, adequate-protein diet. In this study, investigators are going to compare two kinds of the ketogenic diet namely classical ketogenic diet and modified Atkins diet. Fifty children and adolescents with intractable epilepsy will be included, 25 patients in each group, and will receive the diet for three months on non-randomised basis. In the classical ketogenic diet, the diet with a ratio of 4 to 1 (4:1), each 4 grams of fat to each gram of carbohydrate plus protein, will be introduced. Classical ketogenic diet will be established on outpatient setting, without fasting and gradually. The modified Atkins diet will be applied by the ratio of 1:1 or 2:1, each 1 or 2 grams of fat to each gram of carbohydrate plus protein.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents age 1 to 18 years Have not responded well to at least two primary and one secondary antiepileptic drugs Have not received ketogenic diet therapy previously Absence of renal diseases history Absence of cardiovascular diseases history Absence of thyroid function disorders history Absence of cholesterol level more than 300 mg/dl and Triglyceride level more than 200 mg/dl Absence of inherited metabolic disorders that are contraindicated for ketogenic diet therapy including fatty acid oxidation disorders

Exclusion Criteria:

* Onset of complications that threat the life of the patient Inability to continue the diet Unwillingness to adhere the diet

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of the outpatient classical ketogenic diet and modified atkins diet | Prior to and three months after initiation of the classical ketogenic diet and modified Atkins diet

SECONDARY OUTCOMES:
Comparison of the nutritional status of children and adolescents on the classical KD and MAD | Baseline and three months after initiation of the classical ketogenic diet and modified Atkins diet
Comparison of the lipid profiles of children and adolescents on the classical KD and MAD | Baseline and three months after initiation of the classical ketogenic diet and modified Atkins diet
Comparison of the serum electrolytes levels of children and adolescents on the classical KD and MAD | Baseline and three months after initiation of the classical ketogenic diet and modified Atkins diet

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens' Medical Center, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
The IPD would not share with other researchers.